CLINICAL TRIAL: NCT02106390
Title: A Phase 3b, Open-Label, Randomized, Multicenter Study to Assess the Safety and Immunogenicity of GlaxoSmithKline Biologicals Meningococcal Group B Vaccine When Administered Concomitantly With GlaxoSmithKline Biologicals MenACWY Conjugate Vaccine to Healthy Infants
Brief Title: Safety and Immunogenicity of GlaxoSmithKline Biologicals Meningococcal Group B Vaccine When Administered Concomitantly With GlaxoSmithKline Biologicals MenACWY Conjugate Vaccine to Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 205240; V72_56 (Other: Novartis); 2016-005117-44 (EudraCT Number)
Record Dates: First submitted 2014-02-14; First posted 2014-04-08 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-01

CONDITIONS: Infections, Meningococcal
Keywords: Central Nervous System Diseases; Nervous System Diseases; Meningitis
MeSH Terms: conditions — Meningococcal Infections; Central Nervous System Diseases; Nervous System Diseases; Meningitis | interventions — 4CMenB vaccine; MenACWY; Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rMenB+ACWY (Experimental): Approximately 250 healthy infants who will be vaccinated at 3, 5, 7 and 13 months of age.
  Interventions: Biological: Meningococcal group B Vaccine, rMenB+OMV NZ; Biological: Meningococcal ACWY Conjugate Vaccine, MenACWY
- rMENB (Active Comparator): Approximately 250 healthy infants who will be vaccinated at 3, 5, 7 and 13 months of age.
  Interventions: Biological: Meningococcal group B Vaccine, rMenB+OMV NZ
- MenACWY (Active Comparator): Approximately 250 healthy infants who will be vaccinated at 3, 5, 7 and 13 months of age.
  Interventions: Biological: Meningococcal ACWY Conjugate Vaccine, MenACWY

INTERVENTIONS:
Biological: Meningococcal group B Vaccine, rMenB+OMV NZ — 4 doses administered intramuscularly on Days 1, 61, 121 and 301 with blood draw visits at Days 1, 151, 301 and 331 and who will receive reminder calls at 2 and 4 days after each vaccination visit and safety calls on Days 201 and 251.
  Other Names: Bexsero®
  Arms: rMENB; rMenB+ACWY
Biological: Meningococcal ACWY Conjugate Vaccine, MenACWY — 4 doses administered intramuscularly on Days 1, 61, 121 and 301 with blood draw visits at Days 1, 151, 301 and 331 and who will receive reminder calls at 2 and 4 days after each vaccination visit and safety calls on Days 201 and 251.
  Other Names: Menveo®
  Arms: MenACWY; rMenB+ACWY

SUMMARY:
The purpose of this trial is to evaluate the immunogenicity, the safety and the tolerability of rMenB+OMV NZ and MenACWY vaccines in healthy infants, when concomitantly administered at 3, 5, 7 and 13 months of age, compared to either alone.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy 3-month old infants (85-119 days, inclusive) at time of Visit 1 whose parents/legal guardians have given written informed consent after the nature of the study has been explained.
2. Available for all the visits scheduled in the study.
3. In good health as determined by medical history, physical examination and clinical judgment of the investigator.

Exclusion Criteria:

1. History of any previous immunization with a meningococcal vaccine or vaccine containing meningococcal antigen(s) at the time of enrollment.
2. Previous known or suspected disease caused by N. meningitidis.
3. Household contact with and/or intimate exposure to an individual with laboratory confirmed N. meningitidis infection or colonization.
4. History of severe allergic reaction after previous vaccinations, or hypersensitivity to any component of the vaccine.
5. Known or suspected autoimmune disease or impairment/alteration of the immune system resulting from, for ex-ample:

   * Chronic administration of immunosuppressants or other immune-modifying drugs since birth (3 months prior). (For corticosteroids, this means prednisone, or equivalent, ≥ 0.5 mg/kg/day or ≥ 10 mcg/day for children below 2 years. Inhaled and topical steroids are allowed),
   * Immune deficiency disorder, or known HIV infection.
6. Receipt of blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation since birth.
7. History of any progressive or severe neurologic disorder, or seizure disorder or Guillan Barré syndrome (exception: one self-limited febrile seizure is acceptable).
8. History of any bleeding disorder considered as a contraindication to intramuscular injection or blood draw.
9. Child's parent(s) or legal guardian(s) are not able to comprehend and to follow all required study procedures for the whole period of the study.
10. Receipt of any investigational or non-registered product since birth (3 month prior) or are expected to receive during the study period.
11. Family members or household members of site research staff.
12. Any clinically-significant chronic or progressive disease according to judgment of the investigator (pulmonary, cardiovascular, renal, hepatic or endocrine functional abnormality) or a congenital anomaly/known cytogenic disorder (e.g., Down's syndrome).
13. History or any illness/condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study.

Ages: 85 Days to 119 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 750 (Actual)
Dates: Start 2014-06-05 (Actual); Primary Completion 2016-10-14 (Actual); Study Completion 2016-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Argentina (2):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Córdoba
- Mexico (2):
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, Morelia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 750 healthy infants, aged 3 months were recruited from 3 sites in Argentina and 4 sites in Mexico.
Pre-assignment Details: All enrolled subjects were included in the study.
Groups:
- rMenB+ACWY Group: Approximately 250 healthy infants aged 3 months who received 4 doses of rMenB + OMV NZ / MenACWY vaccines, concomitantly administered at 3, 5, 7 and 13 months of age.
- rMenB Group: Approximately 250 healthy infants aged 3 months who received 4 doses of rMenB + OMV NZ administered at 3, 5, 7 and 13 months of age.
- MenACWY Group: Approximately 250 healthy infants aged 3 months who received 4 doses of MenACWY administered at 3, 5, 7 and 13 months of age.
Period: Overall Study
Arm/Group | rMenB+ACWY Group | rMenB Group | MenACWY Group
Started | 252 | 250 | 248
Completed | 203 | 202 | 205
Not Completed | 49 | 48 | 43
Not completed — Withdrawal by Subject | 15 | 16 | 15
Not completed — Lost to Follow-up | 25 | 20 | 13
Not completed — Other: Administrative Reason | 8 | 5 | 12
Not completed — Other: Unspecified | 1 | 4 | 2
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rMenB+ACWY Group | rMenB Group | MenACWY Group | Total
Number analyzed (Participants) | 252 | 250 | 248 | 750
Age, Continuous [Mean (Standard Deviation); unit: Days] | 104.0 (10.72) | 101.4 (10.57) | 102.7 (10.9) | 102.7 (10.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 118 | 139 | 377
  Male | 132 | 132 | 109 | 373
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17 | 20 | 17 | 54
  Other | 235 | 230 | 231 | 696

OUTCOME MEASURES:

1. Primary Outcome: Human Serum Bactericidal Activity (hSBA) Geometric Mean Titers (GMTs) Against Each of the Serogroup B Indicator Strains
Description: Human serum bactericidal activity (hSBA) titers against each of the serogroup B indicator strains-H44/76,5/99,NZ98/254 & M10713 after receiving 4 doses of rMenB+OMV NZ / MenACWY vaccines, concomitantly administered, versus corresponding response in subjects who received rMenB+OMV NZ administered alone, were presented in terms of vaccine group specific geometric mean titers (GMTs).
  This outcome measure applies to only rMenB+ACWY and rMenB groups as the serogroup B indicator strains were assessed only for these two groups.
Time Frame: At Day 331 (one month after the fourth vaccination)
Population: Analysis was performed on the Per Protocol set (PPS). The PPS included all subjects who received a study vaccination and provided an evaluable serum sample at one month after the fourth vaccination and were not excluded due to reasons defined prior to analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | rMenB+ACWY Group | rMenB Group
Number analyzed (Participants) | 148 | 158
Titers
  H44/76: number analyzed (Participants) | 115 | 153
  H44/76 | 92 [67 to 128] | 104 [77 to 141]
  5/99: number analyzed (Participants) | 113 | 148
  5/99 | 1850 [1122 to 3050] | 1790 [1128 to 2842]
  NZ98/254 | 39 [29 to 53] | 38 [28 to 52]
  M10713: number analyzed (Participants) | 131 | 157
  M10713 | 13 [7.82 to 21] | 12 [7.72 to 20]
Statistical Analysis 1: Comparison: rMenB+ACWY Group vs rMenB Group; H44/76- The comparison of adjusted GMTs ratio (rMenB+OMV NZ + MenACWY versus rMenB+OMV NZ) was performed for the H44/76 serogroup B indicator strain,at one month after the fourth vaccination."; Test type: Non-Inferiority — Non-inferiority was to be concluded if, at one month following the fourth vaccination, the lower limits of the two-sided 95% confidence interval for the between-group ratios of GMTs (rMenB+OMV NZ + MenACWY versus rMenB+OMV NZ is > 0.5 for all serogroup B indicator strains; ANOVA; The 2-sided 95% CI for each between groups ratio of GMTs was constructed from an analysis of ANOVA with vaccine group & center as factors in the model; GMT ratio = 0.89, 95% CI 2-sided [0.71 to 1.10]
Statistical Analysis 2: Comparison: rMenB+ACWY Group vs rMenB Group; 5/99-The comparison of adjusted GMTs ratio (rMenB+OMV NZ + MenACWY versus rMenB+OMV NZ) was performed for the 5/99 serogroup B indicator strain,at one month after the fourth vaccination; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; GMT ratio = 1.03, 95% CI 2-sided [0.74 to 1.45]
Statistical Analysis 3: Comparison: rMenB+ACWY Group vs rMenB Group; NZ98/254-The comparison of adjusted GMTs ratio (rMenB+OMV NZ + MenACWY versus rMenB+OMV NZ) was performed for the NZ98/254 serogroup B indicator strain,at one month after the fourth vaccination; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; GMT ratio = 1.01, 95% CI 2-sided [0.82 to 1.25]
Statistical Analysis 4: Comparison: rMenB+ACWY Group vs rMenB Group; M10713-The comparison of adjusted GMTs ratio (rMenB+OMV NZ + MenACWY versus rMenB+OMV NZ) was performed for the M10713 serogroup B indicator strain,at one month after the fourth vaccination; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; GMT ratio = 1.03, 95% CI 2-sided [0.77 to 1.40]

2. Primary Outcome: hSBA Geometric Mean Titers (GMTs) Against Each of the Serogroups A, C, W-135 and Y
Description: hSBA titers against N. meningitidis serogroups A, C, W-135 and Y after receiving four doses of either rMenB+OMV NZ / MenACWY concomitantly administered versus corresponding response in subjects who received MenACWY administered alone were presented in terms of vaccine group specific GMTs.
  This outcome measure applies to only rMenB+ACWY and MenACWY groups as the serogroups A,C,W-135 & Y were assessed only for these two groups.
Time Frame: At Day 331 (one month after the fourth vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | rMenB+ACWY Group | MenACWY Group
Number analyzed (Participants) | 161 | 156
Titers
  Serogroup A: number analyzed (Participants) | 159 | 156
  Serogroup A | 409 [300 to 556] | 165 [122 to 224]
  Serogroup C: number analyzed (Participants) | 157 | 149
  Serogroup C | 452 [312 to 655] | 421 [294 to 602]
  Serogroup W: number analyzed (Participants) | 144 | 143
  Serogroup W | 721 [493 to 1053] | 536 [370 to 776]
  Serogroup Y | 410 [293 to 575] | 391 [280 to 546]
Statistical Analysis 1: Comparison: rMenB+ACWY Group vs MenACWY Group; Serogroup A-The comparison of adjusted GMTs ratio (rMenB+OMV NZ + Men ACWY versus MenACWY) was performed for serogroup A at one month after the fourth vaccination; Test type: Non-Inferiority — Non-inferiority was to be concluded if, at one month following the fourth vaccination, the lower limits of the two-sided 95% confidence interval for the between-group ratios of GMTs (rMenB+OMVNZ + MenACWY versus MenACWY) was > 0.5 for all serogroups A, C, W-135 and Y; ANOVA; [statistical method as in outcome 1, analysis 1]; GMT ratio = 2.48, 95% CI 2-sided [1.97 to 3.11]
Statistical Analysis 2: Comparison: rMenB+ACWY Group vs MenACWY Group; Serogroup C-The comparison of adjusted GMTs ratio (rMenB+OMV NZ + Men ACWY versus MenACWY) was performed for the serogroup C at one month after the fourth vaccination; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; GMT ratio = 1.07, 95% CI 2-sided [0.83 to 1.38]
Statistical Analysis 3: Comparison: rMenB+ACWY Group vs MenACWY Group; Serogroup W-The comparison of adjusted GMTs ratio (rMenB+OMV NZ + Men ACWY versus MenACWY) was performed for the serogroup W-135 at one month after the fourth vaccination; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; GMT ratio = 1.34, 95% CI 2-sided [1.04 to 1.74]
Statistical Analysis 4: Comparison: rMenB+ACWY Group vs MenACWY Group; Serogroup Y-The comparison of adjusted GMTs ratio (rMenB+OMV NZ + Men ACWY versus MenACWY) was performed for the serogroup Y at one month after the fourth vaccination; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; GMT ratio = 1.05, 95% CI 2-sided [0.82 to 1.35]

3. Secondary Outcome: hSBA Geometric Mean Titers Against Each of the Serogroup B Indicator Strains.
Description: hSBA GMTs against each of the N. meningitidis serogroup B indicator strains-H44/76,5/99,NZ98/254 & M10713 at baseline (Day 1).
  This outcome measure applies to only rMenB+ACWY and rMenB groups as the serogroup B strains were assessed only for these two groups.
Time Frame: At Day 1
Population: Analysis was performed on the Full Analysis Set( FAS). The FAS included all subjects who received a study vaccination and provided an evaluable serum sample at baseline (day 1).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | rMenB+ACWY Group | rMenB Group
Number analyzed (Participants) | 191 | 206
Titers
  H44/76: number analyzed (Participants) | 162 | 198
  H44/76 | 1.03 [0.99 to 1.08] | 1.02 [0.98 to 1.07]
  5/99: number analyzed (Participants) | 157 | 192
  5/99 | 1.09 [0.99 to 1.21] | 1.07 [0.97 to 1.17]
  NZ98/254 | 1.06 [1.01 to 1.12] | 1.07 [1.02 to 1.12]
  M10713: number analyzed (Participants) | 182 | 203
  M10713 | 1.88 [1.51 to 2.34] | 1.59 [1.29 to 1.96]

4. Secondary Outcome: hSBA Geometric Mean Titers Against Each of the Serogroup B Indicator Strains.
Description: hSBA GMTs against each of the N. meningitidis serogroup B indicator strains-H44/76,5/99,NZ98/254 & M10713 at one month after the third vaccination (Day 151).
  This outcome measure applies to only rMenB+ACWY and rMenB groups as the serogroup B strains were assessed only for these two groups.
Time Frame: At Day 151 (one month after the third vaccination)
Population: Analysis was performed on the Full Analysis Set( FAS). The FAS included all subjects who received a study vaccination and provided an evaluable serum sample at one month after the third vaccination (Day 151)
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | rMenB+ACWY Group | rMenB Group
Number analyzed (Participants) | 181 | 206
Titers
  H44/76: number analyzed (Participants) | 149 | 199
  H44/76 | 116 [100 to 135] | 129 [113 to 147]
  5/99: number analyzed (Participants) | 137 | 188
  5/99 | 891 [752 to 1055] | 935 [803 to 1088]
  NZ98/254: number analyzed (Participants) | 181 | 205
  NZ98/254 | 32 [26 to 39] | 33 [27 to 40]
  M10713: number analyzed (Participants) | 168 | 206
  M10713 | 9.09 [6.57 to 13] | 10 [7.50 to 14]

5. Secondary Outcome: hSBA Geometric Mean Titers Against Each of the Serogroup B Indicator Strains.
Description: hSBA GMTs against each of the N. meningitidis serogroup B indicator strains-H44/76,5/99,NZ98/254 & M10713 before the fourth vaccination (Day 301).
  This outcome measure applies to only rMenB+ACWY and rMenB groups as the serogroup B strains were assessed only for these two groups.
Time Frame: At Day 301 (before the fourth vaccination)
Population: Analysis was performed on the Full Analysis Set( FAS). The FAS included all subjects who received a study vaccination and provided an evaluable serum sample before the fourth vaccination( Day 301).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | rMenB+ACWY Group | rMenB Group
Number analyzed (Participants) | 173 | 204
Titers
  H44/76: number analyzed (Participants) | 130 | 190
  H44/76 | 7.68 [5.91 to 9.99] | 8.31 [6.54 to 11]
  5/99: number analyzed (Participants) | 139 | 189
  5/99 | 131 [107 to 161] | 109 [90 to 132]
  NZ98/254 | 3.21 [2.44 to 4.21] | 2.93 [2.25 to 3.81]
  M10713: number analyzed (Participants) | 151 | 198
  M10713 | 2.48 [1.89 to 3.27] | 2.40 [1.85 to 3.10]

6. Secondary Outcome: hSBA Geometric Mean Titers Against Each of the Serogroup B Indicator Strains.
Description: hSBA GMTs against each of the N. meningitidis serogroup B indicator strains-H44/76,5/99,NZ98/254 & M10713 at one month after the fourth vaccination (Day 331).
  This outcome measure applies to only rMenB+ACWY and rMenB groups as the serogroup B strains were assessed only for these two groups.
Time Frame: At Day 331 (one month after the fourth vaccination)
Population: Analysis was performed on the Full Analysis Set( FAS). The FAS included all subjects who received a study vaccination and provided an evaluable serum sample at one month after the fourth vaccination( Day 331).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | rMenB+ACWY Group | rMenB Group
Number analyzed (Participants) | 181 | 196
Titers
  H44/76: number analyzed (Participants) | 141 | 188
  H44/76 | 122 [98 to 151] | 126 [104 to 154]
  5/99: number analyzed (Participants) | 143 | 183
  5/99 | 1404 [1016 to 1939] | 1262 [934 to 1706]
  NZ98/254 | 37 [30 to 45] | 36 [30 to 44]
  M10713: number analyzed (Participants) | 161 | 194
  M10713 | 18 [14 to 24] | 17 [13 to 22]

7. Secondary Outcome: hSBA Geometric Mean Titers Against Each of the Serogroups A,C,W-135 & Y.
Description: hSBA GMTs against each of the N. meningitidis serogroups A, C, W-135, Y at baseline (Day 1).
  This outcome measure applies to only rMenB+ACWY and MENACWY groups as the serogroups A,C,W-135 & Y were assessed only for these two groups.
Time Frame: At Day 1
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | rMenB+ACWY Group | MenACWY Group
Number analyzed (Participants) | 213 | 210
Titers
  Serogroup A: number analyzed (Participants) | 211 | 206
  Serogroup A | 2.05 [1.97 to 2.15] | 2.08 [1.99 to 2.17]
  Serogroup C: number analyzed (Participants) | 206 | 204
  Serogroup C | 2.16 [1.98 to 2.35] | 2.09 [1.92 to 2.27]
  Serogroup W: number analyzed (Participants) | 194 | 196
  Serogroup W | 2.33 [2.13 to 2.55] | 2.31 [2.11 to 2.52]
  Serogroup Y | 2.06 [1.95 to 2.17] | 2.16 [2.05 to 2.28]

8. Secondary Outcome: hSBA Geometric Mean Titers Against Each of the Serogroups A, C, W-135 and Y
Description: hSBA GMTs against each of the N. meningitidis serogroups A, C, W-135, Y at one month after the third vaccination (Day 151).
  This outcome measure applies to only rMenB+ACWY and MENACWY groups as the serogroups A,C,W-135 & Y were assessed only for these two groups.
Time Frame: At Day 151 (one month after the third vaccination)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | rMenB+ACWY Group | MenACWY Group
Number analyzed (Participants) | 215 | 214
Titers
  Serogroup A: number analyzed (Participants) | 214 | 210
  Serogroup A | 303 [242 to 379] | 136 [108 to 169]
  Serogroup C: number analyzed (Participants) | 208 | 204
  Serogroup C | 388 [320 to 469] | 416 [345 to 502]
  Serogroup W: number analyzed (Participants) | 178 | 188
  Serogroup W | 347 [282 to 427] | 298 [244 to 364]
  Serogroup Y | 226 [182 to 282] | 283 [228 to 351]

9. Secondary Outcome: hSBA Geometric Mean Titers Against Each of the Serogroups A,C,W-135 & Y.
Description: hSBA GMTs against each of the N. meningitidis serogroups A, C, W-135, Y before the fourth vaccination (Day 301).
  This outcome measure applies to only rMenB+ACWY and MENACWY groups as the serogroups A,C,W-135 & Y were assessed only for these two groups.
Time Frame: At Day 301 (before the fourth vaccination)
Population: Analysis was performed on the Full Analysis Set( FAS). The FAS included all subjects who received a study vaccination and provided an evaluable serum sample before the fourth vaccination(Day 301)
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | rMenB+ACWY Group | MenACWY Group
Number analyzed (Participants) | 203 | 204
Titers
  Serogroup A: number analyzed (Participants) | 200 | 200
  Serogroup A | 20 [15 to 28] | 15 [11 to 21]
  Serogroup C: number analyzed (Participants) | 196 | 189
  Serogroup C | 31 [23 to 41] | 43 [32 to 58]
  Serogroup W: number analyzed (Participants) | 169 | 178
  Serogroup W | 48 [37 to 63] | 47 [36 to 62]
  Serogroup Y | 38 [30 to 49] | 43 [33 to 55]

10. Secondary Outcome: hSBA Geometric Mean Titers Against Each of the Serogroups A,C,W-135 & Y.
Description: hSBA GMTs against each of the N.meningitidis serogroups A, C, W-135, Y at one month after the fourth vaccination (Day 331).
  This outcome measure applies to only rMenB+ACWY and MENACWY groups as the serogroups A,C,W-135 & Y were assessed only for these two groups.
Time Frame: At Day 331 (one month after the fourth vaccination)
Population: Analysis was performed on the Full Analysis Set( FAS). The FAS included all subjects who received a study vaccination and provided an evaluable serum sample at one month after the fourth vaccination (Day 331).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | rMenB+ACWY Group | MenACWY Group
Number analyzed (Participants) | 199 | 204
Titers
  Serogroup A: number analyzed (Participants) | 197 | 203
  Serogroup A | 329 [269 to 403] | 132 [108 to 161]
  Serogroup C: number analyzed (Participants) | 193 | 194
  Serogroup C | 331 [268 to 409] | 311 [252 to 384]
  Serogroup W: number analyzed (Participants) | 179 | 184
  Serogroup W | 576 [458 to 723] | 428 [342 to 537]
  Serogroup Y | 377 [304 to 466] | 363 [294 to 448]

11. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥1:5 Against Each of the Serogroup B Indicator Strains
Description: Percentage of subjects with hSBA titers≥ 1:5 against each of the N. meningitidis serogroup B indicator strains-H44/76,5/99,NZ98/254 & M10713 before the first vaccination (Day 1).
  This outcome measure applies to only rMenB+ACWY and rMenB groups as the serogroup B strains were assessed only for these two groups.
Time Frame: At Day 1
Population: Analysis was performed on the Full Analysis Set( FAS). The FAS included all subjects who received a study vaccination and provided an evaluable serum sample at baseline(Day 1)
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB+ACWY Group | rMenB Group
Number analyzed (Participants) | 191 | 206
Percentage of subjects
  H44/76: number analyzed (Participants) | 162 | 198
  H44/76 | 0 [0.0 to 2.3] | 1 [0.01 to 2.8]
  5/99: number analyzed (Participants) | 157 | 192
  5/99 | 1 [0.15 to 4.5] | 1 [0.13 to 3.7]
  NZ98/254 | 1 [0.01 to 2.9] | 1 [0.01 to 2.7]
  M10713: number analyzed (Participants) | 182 | 203
  M10713 | 16 [11.4 to 22.7] | 11 [6.9 to 15.9]

12. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥1:5 Against Each of the Serogroup B Indicator Strains
Description: Percentage of subjects with hSBA titers ≥ 1:5 against each of the N. meningitidis serogroup B indicator strains-H44/76,5/99,NZ98/254 & M10713 one month after the third vaccination (Day 151).
  This outcome measure applies to only rMenB+ACWY and rMenB groups as the serogroup B indicator strains were assessed only for these two groups.
Time Frame: At Day 151 (one month after the third vaccination)
Population: Analysis was performed on the Full Analysis Set( FAS). The FAS included all subjects who received a study vaccination, provided an evaluable serum sample at one month after the third vaccination (Day 151).
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB+ACWY Group | rMenB Group
Number analyzed (Participants) | 181 | 206
Percentage of subjects
  H44/76: number analyzed (Participants) | 149 | 199
  H44/76 | 100 [97.6 to 100.0] | 100 [98.2 to 100.0]
  5/99: number analyzed (Participants) | 137 | 188
  5/99 | 100 [97.3 to 100.0] | 100 [98.1 to 100.0]
  NZ98/254: number analyzed (Participants) | 181 | 205
  NZ98/254 | 96 [92.2 to 98.4] | 97 [93.7 to 98.9]
  M10713: number analyzed (Participants) | 168 | 206
  M10713 | 70 [62.7 to 77.0] | 68 [61.1 to 74.3]

13. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥1:5 Against Each of the Serogroup B Strains.
Description: Percentage of subjects with hSBA titers ≥ 1:5 against each of the N. meningitidis serogroup B indicator strains-H44/76,5/99,NZ98/254 & M10713 before the fourth vaccination (Day 301).
  This outcome measure applies to only rMenB+ACWY and rMenB groups as the serogroup B indicator strains were assessed only for these two groups.
Time Frame: At Day 301 (before the fourth vaccination)
Population: Analysis was performed on the Full Analysis Set( FAS). The FAS included all subjects who received a study vaccination, provided an evaluable serum sample before the fourth vaccination(Day 301).
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB+ACWY Group | rMenB Group
Number analyzed (Participants) | 173 | 204
Percentage of subjects
  H44/76: number analyzed (Participants) | 130 | 190
  H44/76 | 74 [65.4 to 81.2] | 75 [67.9 to 80.7]
  5/99: number analyzed (Participants) | 139 | 189
  5/99 | 100 [97.4 to 100.0] | 97 [93.9 to 99.1]
  NZ98/254 | 42 [34.2 to 49.3] | 36 [29.7 to 43.3]
  M10713: number analyzed (Participants) | 151 | 198
  M10713 | 33 [25.7 to 41.2] | 31 [24.5 to 37.7]

14. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥1:5 Against Each of the Serogroup B Strains.
Description: Percentage of subjects with hSBA titers ≥ 1:5 against each of the N. meningitidis serogroup B indicator strains-H44/76,5/99,NZ98/254 & M10713 one month after the fourth vaccination (Day 331).
  This outcome measure applies to only rMenB+ACWY and rMenB groups as the serogroup B indicator strains were assessed only for these two groups.
Time Frame: At Day 331 (One month after the fourth vaccination)
Population: Analysis was performed on the Full Analysis Set( FAS). The FAS included all subjects who received a study vaccination, provided an evaluable serum sample at one month after the fourth vaccination (Day 331)
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB+ACWY Group | rMenB Group
Number analyzed (Participants) | 181 | 196
Percentage of subjects
  H44/76: number analyzed (Participants) | 141 | 188
  H44/76 | 100 [97.4 to 100.0] | 99 [97.1 to 99.99]
  5/99: number analyzed (Participants) | 143 | 183
  5/99 | 99 [95.0 to 99.83] | 97 [93.0 to 98.8]
  NZ98/254 | 100 [98.0 to 100.0] | 98 [94.9 to 99.4]
  M10713: number analyzed (Participants) | 161 | 194
  M10713 | 87 [80.8 to 91.7] | 87 [81.6 to 91.5]

15. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥1:8 Against Each of the Serogroup B Indicator Strains
Description: Percentage of subjects with hSBA titers ≥ 1:8 against each of the N. meningitidis serogroup B indicator strains at baseline (Day 1).
  This outcome measure applies to only rMenB+ACWY and rMenB groups as the serogroup B indicator strains were assessed only for these two groups.
Time Frame: At Day 1
Population: Analysis was performed on the Full Analysis Set( FAS). The FAS included all subjects who received a study vaccination, provided an evaluable serum sample at baseline (day 1)
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB+ACWY Group | rMenB Group
Number analyzed (Participants) | 191 | 206
Percentage of subjects
  H44/76: number analyzed (Participants) | 162 | 198
  H44/76 | 0 [0.0 to 2.3] | 0 [0.0 to 1.8]
  5/99: number analyzed (Participants) | 157 | 192
  5/99 | 1 [0.02 to 3.5] | 1 [0.01 to 2.9]
  NZ98/254 | 1 [0.01 to 2.9] | 1 [0.01 to 2.7]
  M10713: number analyzed (Participants) | 182 | 203
  M10713 | 12 [7.3 to 17.1] | 8 [4.6 to 12.5]

16. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥1:8 Against Each of the Serogroup B Indicator Strains
Description: Percentage of subjects with hSBA titers ≥ 1:8 against each of the N. meningitidis serogroup B indicator strains at one month after third vaccination (Day 151).
  This outcome measure applies to only rMenB+ACWY and rMenB groups as the serogroup B indicator strains were assessed only for these two groups.
Time Frame: At Day 151 (one month after the third vaccination)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB+ACWY Group | rMenB Group
Number analyzed (Participants) | 181 | 206
Percentage of subjects
  H44/76: number analyzed (Participants) | 149 | 199
  H44/76 | 100 [97.6 to 100.0] | 100 [98.2 to 100.0]
  5/99: number analyzed (Participants) | 137 | 188
  5/99 | 100 [97.3 to 100.0] | 100 [98.1 to 100.0]
  NZ98/254: number analyzed (Participants) | 181 | 205
  NZ98/254 | 92 [87.4 to 95.7] | 92 [87.6 to 95.5]
  M10713: number analyzed (Participants) | 168 | 206
  M10713 | 65 [57.2 to 72.1] | 59 [52.2 to 66.0]

17. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥1:8 Against Each of the Serogroup B Indicator Strains
Description: Percentage of subjects with hSBA titers ≥ 1:8 against each of the N. meningitidis serogroup B indicator strains before the fourth vaccination (Day 301).
  This outcome measure applies to only rMenB+ACWY and rMenB groups as the serogroup B indicator strains were assessed only for these two groups.
Time Frame: At Day 301 (before the fourth vaccination)
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB+ACWY Group | rMenB Group
Number analyzed (Participants) | 173 | 204
Percentage of subjects
  H44/76: number analyzed (Participants) | 130 | 190
  H44/76 | 58 [49.5 to 67.0] | 56 [48.9 to 63.5]
  5/99: number analyzed (Participants) | 139 | 189
  5/99 | 100 [97.4 to 100.0] | 97 [93.2 to 98.8]
  NZ98/254 | 26 [19.6 to 33.2] | 26 [20.6 to 33.1]
  M10713: number analyzed (Participants) | 151 | 198
  M10713 | 21 [14.4 to 27.9] | 23 [17.5 to 29.7]

18. Secondary Outcome: Percentage of Subjects With hSBA Titers≥1:8 Against Each of the Serogroup B Indicator Strains
Description: Percentage of subjects with hSBA titers≥ 1:8 against each of the N. meningitidis serogroup B indicator strains-H44/76,5/99,NZ98/254 & M10713 at one month after the fourth vaccination (Day 331).
  This outcome measure applies to only rMenB+ACWY and rMenB groups as the serogroup B indicator strains were assessed only for these two groups.
Time Frame: At Day 331 (one month after the fourth vaccination)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB+ACWY Group | rMenB Group
Number analyzed (Participants) | 181 | 196
Percentage of subjects
  H44/76: number analyzed (Participants) | 141 | 188
  H44/76 | 100 [97.4 to 100.0] | 99 [97.1 to 99.99]
  5/99: number analyzed (Participants) | 143 | 183
  5/99 | 99 [95.0 to 99.83] | 97 [93.0 to 98.8]
  NZ98/254 | 98 [94.4 to 99.4] | 94 [90.2 to 97.2]
  M10713: number analyzed (Participants) | 161 | 194
  M10713 | 83 [76.5 to 88.6] | 82 [76.4 to 87.5]

19. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥1:4 Against Each of the Serogroups A, C, W-135 and Y
Description: Percentage of subjects with hSBA titers≥ 1:4 against each of the N. meningitidis serogroups A, C, W-135 and Y before the first vaccination (Day 1).
  This outcome measure applies to only rMenB+ACWY and MENACWY groups as the serogroups were assessed only for these two groups.
Time Frame: At Day 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB+ACWY Group | MenACWY Group
Number analyzed (Participants) | 213 | 210
Percentage of subjects
  Serogroup A: number analyzed (Participants) | 211 | 206
  Serogroup A | 1 [0.11 to 3.4] | 1 [0.12 to 3.5]
  Serogroup C: number analyzed (Participants) | 206 | 204
  Serogroup C | 4 [1.7 to 7.5] | 3 [1.4 to 6.9]
  Serogroup W: number analyzed (Participants) | 194 | 196
  Serogroup W | 4 [1.8 to 8.0] | 4 [1.4 to 7.2]
  Serogroup Y | 2 [0.5 to 4.7] | 5 [2.3 to 8.6]

20. Secondary Outcome: Percentage of Subjects With hSBA Titers≥1:4 Against Each of the Serogroups A, C, W-135 and Y
Description: Percentage of subjects with hSBA titers≥ 1:4 against each of the N. meningitidis serogroups A, C, W-135 and Y at one month after the third vaccination (Day 151). This outcome measure applies to only rMenB+ACWY and MENACWY groups as the serogroups were assessed only for these two groups.
Time Frame: At Day 151 (one month after the third vaccination)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB+ACWY Group | MenACWY Group
Number analyzed (Participants) | 215 | 214
Percentage of subjects
  Serogroup A: number analyzed (Participants) | 214 | 210
  Serogroup A | 99 [97.4 to 99.99] | 96 [92.0 to 98.0]
  Serogroup C: number analyzed (Participants) | 208 | 204
  Serogroup C | 100 [98.2 to 100.0] | 100 [98.2 to 100.0]
  Serogroup W: number analyzed (Participants) | 178 | 188
  Serogroup W | 100 [97.9 to 100.0] | 100 [98.1 to 100.0]
  Serogroup Y | 99 [96.0 to 99.71] | 100 [98.3 to 100.0]

21. Secondary Outcome: Percentage of Subjects With hSBA Titers≥1:4 Against Each of the Serogroups A, C, W-135 and Y
Description: Percentage of subjects with hSBA titers≥ 1:4 against each of the N. meningitidis serogroups A, C, W-135 and Y before the fourth vaccination (Day 301).
  This outcome measure applies to only rMenB+ACWY and MENACWY groups as the serogroups were assessed only for these two groups.
Time Frame: At Day 301 (before the fourth vaccination)
Population: Analysis was performed on the Full Analysis Set( FAS). The FAS included all subjects who received a study vaccination, provided an evaluable serum sample before the fourth vaccination (Day 301).
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB+ACWY Group | MenACWY Group
Number analyzed (Participants) | 203 | 204
Percentage of subjects
  Serogroup A: number analyzed (Participants) | 200 | 200
  Serogroup A | 68 [60.5 to 73.9] | 63 [55.4 to 69.2]
  Serogroup C: number analyzed (Participants) | 196 | 189
  Serogroup C | 88 [82.3 to 92.0] | 89 [84.1 to 93.4]
  Serogroup W: number analyzed (Participants) | 169 | 178
  Serogroup W | 93 [88.7 to 96.7] | 96 [91.3 to 98.0]
  Serogroup Y | 91 [85.8 to 94.3] | 95 [90.6 to 97.3]

22. Secondary Outcome: Percentage of Subjects With hSBA Titers≥1:4 Against Each of the Serogroups A, C, W-135 and Y
Description: Percentage of subjects with hSBA titers≥ 1:4 against each of the N. meningitidis serogroups A, C, W-135 and Y at one month after the fourth vaccination (Day 331). This outcome measure applies to only rMenB+ACWY and MENACWY groups as the serogroups were assessed only for these two groups.
Time Frame: At Day 331 (one month after the fourth vaccination)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB+ACWY Group | MenACWY Group
Number analyzed (Participants) | 199 | 204
Percentage of subjects
  Serogroup A: number analyzed (Participants) | 197 | 203
  Serogroup A | 100 [98.1 to 100.0] | 98 [94.3 to 99.2]
  Serogroup C: number analyzed (Participants) | 193 | 194
  Serogroup C | 100 [98.1 to 100.0] | 100 [98.1 to 100.0]
  Serogroup W: number analyzed (Participants) | 179 | 184
  Serogroup W | 100 [98.0 to 100.0] | 100 [98.0 to 100.0]
  Serogroup Y | 100 [98.2 to 100.0] | 99 [97.3 to 99.99]

23. Secondary Outcome: Within-subject Geometric Mean Ratios (GMRs) Against Each of the Serogroup B Indicator Strains
Description: Geometric Mean Ratios(GMRs) of GMTs against each of the serogroup B indicator strains- H44/76, 5/99, N98/254 & M10713 were calculated at one month after the fourth vaccination (Day 331) versus pre fourth vaccination(Day 301).
Time Frame: At Day 331 (one month after fourth vaccination)
Population: Analysis was performed on the Full Analysis Set( FAS). The FAS included all subjects who received a study vaccination, provided an evaluable serum sample at one month after the fourth vaccination (Day 331) and before the fourth vaccination( Day 301).
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | rMenB+ACWY Group | rMenB Group
Number analyzed (Participants) | 155 | 195
Ratio
  H44/76: number analyzed (Participants) | 109 | 178
  H44/76 | 17 [13 to 22] | 16 [12 to 20]
  5/99: number analyzed (Participants) | 118 | 169
  5/99 | 9.60 [6.99 to 13] | 12 [8.86 to 16]
  NZ98/254 | 11 [8.35 to 15] | 12 [9.39 to 16]
  M10713: number analyzed (Participants) | 130 | 187
  M10713 | 5.99 [4.20 to 8.54] | 6.75 [4.90 to 9.29]

24. Secondary Outcome: Within-subject Geometric Mean Ratios (GMRs) Against Each of Serogroups A, C, W-135 and Y
Description: Geometric Mean Ratios(GMRs) of GMTs against each of the serogroups A,C,W-135 & Y were calculated at one month after the fourth vaccination (Day 331) versus pre fourth vaccination (Day 301).
Time Frame: At Day 331 (one month after the fourth vaccination)
Population: as for outcome 23
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- MenACWY Group: Approximately 250 healthy infants aged 3 months who received 4 doses of rMenB + OMV NZ administered at 3, 5, 7 and 13 months of age.
Arm/Group | rMenB+ACWY Group | MenACWY Group
Number analyzed (Participants) | 197 | 201
Ratio
  Serogroup A: number analyzed (Participants) | 192 | 196
  Serogroup A | 16 [13 to 21] | 8.75 [6.69 to 11]
  Serogroup C: number analyzed (Participants) | 185 | 178
  Serogroup C | 11 [8.86 to 14] | 7.79 [6.25 to 9.71]
  Serogroup W: number analyzed (Participants) | 155 | 161
  Serogroup W | 13 [10 to 16] | 9.44 [7.52 to 12]
  Serogroup Y | 9.75 [8.00 to 12] | 8.97 [7.36 to 11]

25. Secondary Outcome: Percentage of Subjects With Four-fold Increases in hSBA Titers Against Each of the Serogroup B Indicator Strains
Description: Percentage of subjects with four-fold increase in hSBA titers against each of the N. meningitidis serogroup B indicator strains-H44/76,5/99,NZ98/254 & M10713 at one month after the fourth vaccination (Day 331) over pre-fourth vaccination (Day 301).
  This outcome measure applies to only groups rMenB+ACWY and rMenB as the serogroup B indicator strains were assessed only for these two groups.
  For serogroup B strains, 4-fold increase in titers was defined as post 4th vaccination titer ≥8 (if pre 4th vaccination titer was <2) or post 4th vaccination titer ≥ 4 x pre 4th vaccination titer (if pre 4th vaccination titer was ≥2).
Time Frame: At Day 331 (one month after the fourth vaccination)
Population: Analysis was performed on the Full Analysis Set( FAS). The FAS included all subjects who received a study vaccination, provided an evaluable serum sample at one month after the fourth vaccination (Day 331) and before the fourth vaccination (Day 301).
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB+ACWY Group | rMenB Group
Number analyzed (Participants) | 155 | 195
Percentage of subjects
  H44/76: number analyzed (Participants) | 109 | 178
  H44/76 | 93 [86.0 to 96.8] | 92 [87.2 to 95.6]
  5/99: number analyzed (Participants) | 118 | 169
  5/99 | 94 [88.2 to 97.6] | 95 [90.9 to 97.9]
  NZ98/254 | 81 [73.5 to 86.5] | 79 [73.1 to 84.9]
  M10713: number analyzed (Participants) | 130 | 187
  M10713 | 58 [48.7 to 66.3] | 60 [52.5 to 67.0]

26. Secondary Outcome: Percentage of Subjects With Four-fold Increases in hSBA Titers Against Each of the Serogroups A, C, W-135 and Y
Description: Percentages of subjects with four-fold increases in hSBA against each of the N. meningitidis serogroups A,C,W & Y at one month after the fourth vaccination (Day 331) over pre-fourth vaccination(Day 301).
  This outcome measure applies to only rMenB+ACWY and MENACWY groups as the serogroups were assessed only for these two groups.
  For serogroups A, C, W and Y, 4-fold increase in titers was defined as post 4th vaccination titer ≥16 (if pre 4th vaccination titer was <4) or post 4th vaccination titer ≥ 4 x pre 4th vaccination titer (if pre 4th vaccination titer was ≥4).
Time Frame: At Day 331 (one month after the fourth vaccination)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB+ACWY Group | MenACWY Group
Number analyzed (Participants) | 197 | 201
Percentage of subjects
  Serogroup A: number analyzed (Participants) | 192 | 196
  Serogroup A | 90 [84.4 to 93.5] | 71 [64.6 to 77.6]
  Serogroup C: number analyzed (Participants) | 185 | 178
  Serogroup C | 88 [81.9 to 92.0] | 77 [70.1 to 82.9]
  Serogroup W: number analyzed (Participants) | 155 | 161
  Serogroup W | 89 [83.0 to 93.5] | 84 [77.9 to 89.7]
  Serogroup Y | 82 [75.6 to 86.9] | 81 [74.4 to 85.8]

27. Secondary Outcome: Percentage of Subjects With hSBA Titers≥1:8 Against Each of the Serogroups A, C, W-135 and Y
Description: Percentage of subjects with hSBA titers≥ 1:8 against each of the N. meningitidis serogroups A, C, W-135 and Y at baseline (Day 1).
  This outcome measure applies to only rMenB+ACWY and MENACWY groups as the serogroups were assessed only for these two groups.
Time Frame: At Day 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB+ACWY Group | MenACWY Group
Number analyzed (Participants) | 213 | 210
Percentage of subjects
  Serogroup A: number analyzed (Participants) | 211 | 206
  Serogroup A | 1 [0.01 to 2.6] | 1 [0.01 to 2.7]
  Serogroup C: number analyzed (Participants) | 206 | 204
  Serogroup C | 2 [0.8 to 5.6] | 2 [0.5 to 4.9]
  Serogroup W: number analyzed (Participants) | 194 | 196
  Serogroup W | 4 [1.5 to 7.3] | 3 [0.8 to 5.9]
  Serogroup Y | 0 [0.0 to 1.7] | 2 [0.5 to 4.8]

28. Secondary Outcome: Percentage of Subjects With hSBA Titers≥1:8 Against Each of the Serogroups A, C, W-135 and Y
Description: Percentage of subjects with hSBA titers≥ 1:8 against each of the N. meningitidis serogroups A, C, W-135 & Y at one month after the third vaccination (Day 151).
  This outcome measure applies to only rMenB+ACWY and MENACWY groups as the serogroups were assessed only for these two groups.
Time Frame: At Day 151 (one month before the third vaccination)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB+ACWY Group | MenACWY Group
Number analyzed (Participants) | 215 | 214
Percentage of subjects
  Serogroup A: number analyzed (Participants) | 214 | 210
  Serogroup A | 99 [97.4 to 99.99] | 96 [92.0 to 98.0]
  Serogroup C: number analyzed (Participants) | 208 | 204
  Serogroup C | 100 [98.2 to 100.0] | 100 [98.2 to 100.0]
  Serogroup W: number analyzed (Participants) | 178 | 188
  Serogroup W | 100 [97.9 to 100.0] | 99 [97.1 to 99.99]
  Serogroup Y | 98 [95.3 to 99.5] | 99 [97.4 to 99.99]

29. Secondary Outcome: Percentage of Subjects With hSBA Titers≥1:8 Against Each of the Serogroups A, C, W-135 and Y
Description: Percentage of subjects with hSBA titers≥ 1:8 against each of the N. meningitidis serogroups A, C, W-135 & Y before the fourth vaccination (Day 301). This outcome measure applies to only rMenB+ACWY and MENACWY groups as the serogroups were assessed only for these two groups.
Time Frame: At Day 301 (before the fourth vaccination)
Population: Analysis was performed on the Full Analysis Set( FAS). The FAS included all subjects who received a study vaccination and provided an evaluable serum sample before the fourth vaccination (Day 301).
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB+ACWY Group | MenACWY Group
Number analyzed (Participants) | 203 | 204
Percentage of subjects
  Serogroup A: number analyzed (Participants) | 200 | 200
  Serogroup A | 65 [58.0 to 71.6] | 58 [50.8 to 64.9]
  Serogroup C: number analyzed (Participants) | 196 | 189
  Serogroup C | 77 [70.5 to 82.7] | 85 [79.3 to 89.9]
  Serogroup W: number analyzed (Participants) | 169 | 178
  Serogroup W | 92 [86.5 to 95.4] | 91 [85.8 to 94.8]
  Serogroup Y | 86 [80.1 to 90.2] | 91 [85.8 to 94.3]

30. Secondary Outcome: Percentage of Subjects With hSBA Titers≥1:8 Against Each of the Serogroups A, C, W-135 and Y
Description: Percentage of subjects with hSBA titers≥ 1:8 against each of the N. meningitidis serogroups A, C, W-135 & Y at one month after the fourth vaccination (Day 331).
  This outcome measure applies to only rMenB+ACWY and MENACWY groups as the serogroups were assessed only for these two groups.
Time Frame: At Day 331 (one month after the fourth vaccination)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB+ACWY Group | MenACWY Group
Number analyzed (Participants) | 199 | 204
Percentage of subjects
  Serogroup A: number analyzed (Participants) | 197 | 203
  Serogroup A | 100 [98.1 to 100.0] | 96 [92.4 to 98.3]
  Serogroup C: number analyzed (Participants) | 193 | 194
  Serogroup C | 99 [97.1 to 99.99] | 100 [98.1 to 100.0]
  Serogroup W: number analyzed (Participants) | 179 | 184
  Serogroup W | 100 [98.0 to 100.0] | 100 [98.0 to 100.0]
  Serogroup Y | 98 [95.7 to 99.69] | 99 [97.3 to 99.99]

31. Secondary Outcome: Number of Subjects With Solicited Local and Systemic Adverse Events (AEs)
Description: Number of subjects with solicited local and systemic AEs during the 7 days (including the day of vaccination) after any vaccination
Time Frame: From Day 1 (6 hours) to Day 7 after each vaccination (Days 1, 61, 121 and 301)
Population: Analysis was performed on the Solicited Safety Set. The solicited safety set included all subjects who provide informed consent & provide demographic and/or baseline screening assessments, regardless of the subject's randomization and treatment status in the trial and received a subject ID and provided post vaccination solicited adverse events data
Measure: Count of Participants; unit: Participants
Arm/Group | rMenB+ACWY Group | rMenB Group | MenACWY Group
Number analyzed (Participants) | 240 | 232 | 237
Participants
  Any | 235 | 226 | 194
  Any local | 220 | 214 | 157
  Any Systemic | 217 | 217 | 178
  Erythema (vaccination 1): number analyzed (Participants) | 239 | 227 | 232
  Erythema (vaccination 1) | 101 | 102 | 44
  Induration (vaccination 1): number analyzed (Participants) | 239 | 230 | 233
  Induration (vaccination 1) | 111 | 102 | 22
  Swelling (vaccination 1): number analyzed (Participants) | 239 | 229 | 233
  Swelling (vaccination 1) | 82 | 86 | 22
  Tenderness (vaccination 1): number analyzed (Participants) | 239 | 227 | 234
  Tenderness (vaccination 1) | 162 | 159 | 73
  Change in Eating Habits (vaccination 1): number analyzed (Participants) | 238 | 227 | 232
  Change in Eating Habits (vaccination 1) | 53 | 47 | 34
  Diarrhea (vaccination 1): number analyzed (Participants) | 237 | 228 | 234
  Diarrhea (vaccination 1) | 46 | 41 | 42
  Irritability (vaccination 1): number analyzed (Participants) | 237 | 226 | 233
  Irritability (vaccination 1) | 111 | 121 | 87
  Persistent Crying (vaccination 1): number analyzed (Participants) | 237 | 228 | 234
  Persistent Crying (vaccination 1) | 124 | 132 | 85
  Rash (vaccination 1): number analyzed (Participants) | 237 | 225 | 233
  Rash (vaccination 1) | 19 | 28 | 18
  Sleepiness (vaccination 1): number analyzed (Participants) | 238 | 225 | 232
  Sleepiness (vaccination 1) | 69 | 78 | 54
  Vomiting (vaccination 1): number analyzed (Participants) | 237 | 228 | 234
  Vomiting (vaccination 1) | 14 | 28 | 23
  Fever (vaccination 1): number analyzed (Participants) | 239 | 229 | 233
  Fever (vaccination 1) | 49 | 54 | 10
  Treatment of Pain/Fever (vaccination 1): number analyzed (Participants) | 237 | 228 | 227
  Treatment of Pain/Fever (vaccination 1) | 82 | 98 | 25
  Erythema (vaccination 2): number analyzed (Participants) | 227 | 220 | 229
  Erythema (vaccination 2) | 97 | 102 | 47
  Induration (vaccination 2): number analyzed (Participants) | 227 | 221 | 229
  Induration (vaccination 2) | 99 | 110 | 32
  Swelling (vaccination 2): number analyzed (Participants) | 227 | 220 | 229
  Swelling (vaccination 2) | 78 | 83 | 24
  Tenderness (vaccination 2): number analyzed (Participants) | 227 | 221 | 229
  Tenderness (vaccination 2) | 142 | 138 | 66
  Change in Eating Habits (vaccination 2): number analyzed (Participants) | 226 | 220 | 229
  Change in Eating Habits (vaccination 2) | 46 | 44 | 31
  Diarrhea (vaccination 2): number analyzed (Participants) | 226 | 220 | 228
  Diarrhea (vaccination 2) | 37 | 36 | 24
  Irritability (vaccination 2): number analyzed (Participants) | 226 | 220 | 228
  Irritability (vaccination 2) | 99 | 95 | 70
  Persistent Crying (vaccination 2): number analyzed (Participants) | 226 | 220 | 228
  Persistent Crying (vaccination 2) | 104 | 108 | 66
  Rash (vaccination 2): number analyzed (Participants) | 226 | 219 | 228
  Rash (vaccination 2) | 16 | 21 | 13
  Sleepiness (vaccination 2): number analyzed (Participants) | 225 | 220 | 227
  Sleepiness (vaccination 2) | 51 | 55 | 45
  Vomiting (vaccination 2): number analyzed (Participants) | 226 | 220 | 229
  Vomiting (vaccination 2) | 10 | 21 | 17
  Fever (vaccination 2): number analyzed (Participants) | 227 | 218 | 227
  Fever (vaccination 2) | 48 | 54 | 15
  Treatment of Pain/Fever (vaccination 2): number analyzed (Participants) | 226 | 219 | 228
  Treatment of Pain/Fever (vaccination 2) | 74 | 91 | 29
  Erythema (vaccination 3): number analyzed (Participants) | 218 | 215 | 220
  Erythema (vaccination 3) | 86 | 96 | 35
  Induration (vaccination 3): number analyzed (Participants) | 217 | 215 | 221
  Induration (vaccination 3) | 92 | 103 | 30
  Swelling (vaccination 3): number analyzed (Participants) | 218 | 214 | 220
  Swelling (vaccination 3) | 73 | 82 | 19
  Tenderness (vaccination 3): number analyzed (Participants) | 218 | 215 | 222
  Tenderness (vaccination 3) | 139 | 128 | 59
  Change in Eating Habits (vaccination 3): number analyzed (Participants) | 218 | 215 | 221
  Change in Eating Habits (vaccination 3) | 42 | 45 | 33
  Diarrhea (vaccination 3): number analyzed (Participants) | 218 | 215 | 221
  Diarrhea (vaccination 3) | 24 | 40 | 25
  Irritability (vaccination 3): number analyzed (Participants) | 218 | 215 | 220
  Irritability (vaccination 3) | 83 | 84 | 61
  Persistent Crying (vaccination 3): number analyzed (Participants) | 218 | 214 | 221
  Persistent Crying (vaccination 3) | 90 | 92 | 60
  Rash (vaccination 3): number analyzed (Participants) | 218 | 215 | 220
  Rash (vaccination 3) | 10 | 11 | 11
  Sleepiness (vaccination 3): number analyzed (Participants) | 218 | 215 | 221
  Sleepiness (vaccination 3) | 39 | 46 | 39
  Vomiting (vaccination 3): number analyzed (Participants) | 218 | 215 | 221
  Vomiting (vaccination 3) | 7 | 27 | 14
  Fever (vaccination 3): number analyzed (Participants) | 218 | 214 | 222
  Fever (vaccination 3) | 37 | 38 | 25
  Treatment of Pain/Fever (vaccination 3): number analyzed (Participants) | 217 | 215 | 222
  Treatment of Pain/Fever (vaccination 3) | 57 | 69 | 31
  Erythema (vaccination 4): number analyzed (Participants) | 203 | 199 | 204
  Erythema (vaccination 4) | 73 | 88 | 37
  Induration (vaccination 4): number analyzed (Participants) | 203 | 200 | 204
  Induration (vaccination 4) | 84 | 93 | 29
  Swelling (vaccination 4): number analyzed (Participants) | 203 | 200 | 204
  Swelling (vaccination 4) | 75 | 74 | 21
  Tenderness (vaccination 4): number analyzed (Participants) | 203 | 200 | 204
  Tenderness (vaccination 4) | 126 | 129 | 64
  Change in Eating Habits (vaccination 4): number analyzed (Participants) | 203 | 200 | 204
  Change in Eating Habits (vaccination 4) | 59 | 45 | 40
  Diarrhea (vaccination 4): number analyzed (Participants) | 203 | 200 | 204
  Diarrhea (vaccination 4) | 29 | 28 | 23
  Irritability (vaccination 4): number analyzed (Participants) | 203 | 200 | 204
  Irritability (vaccination 4) | 81 | 74 | 57
  Persistent Crying (vaccination 4): number analyzed (Participants) | 203 | 200 | 204
  Persistent Crying (vaccination 4) | 84 | 89 | 56
  Rash (vaccination 4): number analyzed (Participants) | 203 | 200 | 204
  Rash (vaccination 4) | 11 | 13 | 6
  Sleepiness (vaccination 4): number analyzed (Participants) | 203 | 200 | 204
  Sleepiness (vaccination 4) | 50 | 37 | 33
  Vomiting (vaccination 4): number analyzed (Participants) | 203 | 200 | 204
  Vomiting (vaccination 4) | 15 | 14 | 11
  Fever (vaccination 4): number analyzed (Participants) | 203 | 200 | 202
  Fever (vaccination 4) | 53 | 46 | 19
  Treatment of Pain/Fever (vaccination 4): number analyzed (Participants) | 202 | 200 | 204
  Treatment of Pain/Fever (vaccination 4) | 71 | 67 | 31

32. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events
Description: An unsolicited adverse event (AE) is defined as any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product at any dose that does not necessarily have to have a causal relationship with this treatment.
Time Frame: From Day 1 to Day 7 after each vaccination (Days 1, 61, 121 and 301)
Population: Analysis was performed on the Unsolicited Safety Set. The Unsolicited safety set included all subjects who provided informed consent & demographic and/or baseline screening assessments, regardless of the subject's randomization and treatment status in the trial and received a subject ID and provided post-vaccination unsolicited adverse event record
Measure: Count of Participants; unit: Participants
Arm/Group | rMenB+ACWY Group | rMenB Group | MenACWY Group
Number analyzed (Participants) | 249 | 249 | 246
Participants
  Any | 103 | 116 | 70
  Any unsolicited AEs( vaccination 1): number analyzed (Participants) | 240 | 233 | 235
  Any unsolicited AEs( vaccination 1) | 63 | 62 | 20
  Any unsolicited AEs( vaccination 2): number analyzed (Participants) | 230 | 222 | 229
  Any unsolicited AEs( vaccination 2) | 60 | 69 | 29
  Any unsolicited AEs( vaccination 3): number analyzed (Participants) | 220 | 216 | 223
  Any unsolicited AEs( vaccination 3) | 57 | 63 | 23
  Any unsolicited AEs( vaccination 4): number analyzed (Participants) | 203 | 202 | 205
  Any unsolicited AEs( vaccination 4) | 44 | 58 | 13

33. Secondary Outcome: Number of Subjects With SAEs, AEs Leading to Withdrawal and Medically Attended AEs (MAEs)
Description: A serious adverse event is any untoward medical occurrence that at any dose results in death/ is life threatening/requires prolonged hospitalization/Persistent or significant disability/incapacity/congenital anomaly/or birth defect.
Time Frame: Throughout the whole study period (from Day 1 upto Day 331)
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | rMenB+ACWY Group | rMenB Group | MenACWY Group
Number analyzed (Participants) | 249 | 249 | 246
Participants
  Any SAEs | 6 | 13 | 11
  Any Medically Attended AEs | 177 | 188 | 183
  Any AEs leading to premature withdrawal | 0 | 2 | 1

ADVERSE EVENTS:
Time Frame: Solicited local and systemic AEs were collected from day 1 (6 hours) upto day 7 after each vaccination. Unsolicited AEs were collected from day 1 to day 7.
Description: Serious Adverse Events (SAEs) were collected throughout the whole study period (from day 1 to day 331).
  All the unsolicited AEs were reported by non-systematic assessment and the solicited AEs were reported by systematic assessment.
  Out of the 750 subjects enrolled in the study, a total of 744 subjects were exposed to the study vaccine and were included in the overall safety set. Therefore, the number of subjects reporting adverse events are lesser than the number of subjects enrolled.
Arm/Group | rMenB+ACWY Group | rMenB Group | MenACWY Group
All-Cause Mortality (participants affected / at risk) | 0/249 | 0/249 | 0/246
Serious Adverse Events (participants affected / at risk) | 6/249 | 13/249 | 11/246
Other Adverse Events (participants affected / at risk) | 240/249 | 232/249 | 221/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rMenB+ACWY Group (N=249) | rMenB Group (N=249) | MenACWY Group (N=246)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Milk allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 3 (3) | 4 (5)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Exanthema subitum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Kawasaki's disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rMenB+ACWY Group (N=249) | rMenB Group (N=249) | MenACWY Group (N=246)
Diarrhoea (Gastrointestinal disorders) | 108 (181) | 98 (196) | 89 (163)
Vomiting (Gastrointestinal disorders) | 36 (51) | 64 (105) | 49 (82)
Injection site pain (General disorders) | 212 (593) | 207 (583) | 131 (267)
Crying (General disorders) | 176 (434) | 184 (463) | 129 (301)
Injection site erythema (General disorders) | 147 (424) | 162 (480) | 104 (211)
Injection site induration (General disorders) | 144 (575) | 152 (609) | 57 (116)
Injection site swelling (General disorders) | 130 (380) | 138 (403) | 56 (88)
Pyrexia (General disorders) | 125 (201) | 121 (210) | 60 (79)
Nasopharyngitis (Infections and infestations) | 81 (161) | 87 (164) | 78 (135)
Viral upper respiratory tract infection (Infections and infestations) | 72 (104) | 82 (127) | 86 (123)
Pharyngitis (Infections and infestations) | 50 (57) | 50 (59) | 50 (60)
Bronchiolitis (Infections and infestations) | 34 (40) | 34 (37) | 37 (37)
Gastroenteritis (Infections and infestations) | 31 (37) | 40 (44) | 38 (43)
Conjunctivitis (Infections and infestations) | 20 (23) | 18 (18) | 24 (25)
Candida nappy rash (Infections and infestations) | 15 (16) | 12 (14) | 6 (6)
Rhinitis (Infections and infestations) | 14 (17) | 13 (16) | 19 (21)
Viral rash (Infections and infestations) | 13 (13) | 14 (14) | 13 (13)
Somnolence (Nervous system disorders) | 106 (226) | 115 (236) | 87 (189)
Irritability (Psychiatric disorders) | 155 (409) | 170 (418) | 125 (320)
Eating disorder (Psychiatric disorders) | 110 (214) | 100 (194) | 85 (162)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 17 (25) | 12 (16) | 15 (26)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 12 (16) | 13 (23)
Rash (Skin and subcutaneous tissue disorders) | 46 (62) | 57 (81) | 42 (62)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 12 (16) | 16 (16) | 14 (15)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 6 (6) | 11 (12) | 17 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.